CLINICAL TRIAL: NCT00211939
Title: CARE-2 (Calcium Acetate (PhosLo®)/Sevelamer(Renagel®) Evaluation Study 2)
Brief Title: CARE-2 (Calcium Acetate [PhosLo®]/Sevelamer[Renagel®] Evaluation Study 2) for Heart Calcification in Dialysis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nabi Biopharmaceuticals (Industry)
Responsible Party: Paul Kessler, MD, Sr. VP, Clinical, Medical & Regulatory Affairs, Nabi Biopharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Nabi 6404
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2008-01-08 (Estimated); Status verified 2007-12

CONDITIONS: Calcinosis; Arteriosclerosis; Hyperparathyroidism, Secondary
Keywords: PhosLo (Calcium acetate); Renagel (sevelamer, polyallylamine HCL); kidney dialysis; hyperphosphatemia; Kidney failure
MeSH Terms: conditions — Calcinosis; Arteriosclerosis; Hyperparathyroidism, Secondary; Hyperphosphatemia; Renal Insufficiency | interventions — calcium acetate; Sevelamer; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): PhosLo + atorvastatin
  Interventions: Drug: calcium acetate; Drug: atorvastatin
- 2 (Active Comparator): Sevelamer + atorvastatin
  Interventions: Drug: sevelamer; Drug: atorvastatin

INTERVENTIONS:
Drug: calcium acetate — 667 mg gelcap, 2-4 t.i.d titrated to serum phosphorus level
  Other Names: PhosLo
  Arms: 1
Drug: sevelamer — 1-3 tablets t.i.d, titrated to serum phosphorus level
  Other Names: Renagel
  Arms: 2
Drug: atorvastatin — 20 mg PO qD (in PhosLo group), or held until D60 (sevelamer group); titrate by LDL levels and liver function tests
  Other Names: Lipitor

SUMMARY:
The purpose of the study is to evaluate the effects of two phosphate binders, PhosLo and sevelamer, on heart calcification in dialysis patients. The study will use a non-invasive technique, electron beam computed tomography (CT) scanning, to measure calcium in the coronary arteries, the aortic valve, and the mitral valve.

DETAILED DESCRIPTION:
Cardiovascular disease is the major cause of death and disability in patients with end-stage renal disease on hemodialysis. It has been hypothesized that ingestion of calcium-based phosphate binders results in net positive calcium balance and vascular calcium deposition. Chertow et al. tested the role of ingested calcium in the progression of cardiovascular calcification in the Treat-To-Goal study (Kidney International 62:245, 2002). They reported that patients treated with calcium-based phosphate binders demonstrated progressive cardiovascular calcification, while patients treated with a calcium-free binder, sevelamer, showed stabilization or improvement in calcification scores. However, the protocol did not prohibit intake of supplemental oral calcium in the sevelamer group, which confounded their ability to accurately test the calcium hypothesis. Moreover, due to the cholesterol sequestering activities of sevelamer, the low-density lipoprotein (LDL) cholesterol was lower among sevelamer-treated patients than the calcium treated patients, resulting in a major imbalance in a cardiovascular risk factor. Lowering LDL level reduces progression of CVC and therefore confounds interpretation of the study. Subsequently, it has been reported in the lay press that patients randomized to sevelamer or calcium-based binders in the Dialysis Clinical Outcomes Revisited (DCOR) study have failed to show a difference in mortality or major secondary endpoints (Suki et al., To be presented American Society of Nephrology November 2005). To circumvent these limitations, the CARE-2 study will test the hypothesis that if LDL levels are lowered to a similar level in calcium acetate and sevelamer-treated patients, there will be no difference in the progression of cardiac calcification. CARE-2 will randomize patients with elevated LDL to calcium acetate or sevelamer. Atorvastatin is added to achieve LDL < 70 mg/dL in both treatment groups. The primary endpoint is change in cardiac calcification scores, determined by electron beam scanning after 1 year. Secondary endpoints include the ability of calcium acetate and sevelamer to control phosphorus and meet NKF-K/DOQI guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Eligible subjects will be male or female patients with end-stage renal disease on maintenance hemodialysis for less than 5 years, with elevated LDL cholesterol
* Currently treated with oral phosphate binders
* Coronary artery calcium scores of 30 to 5000 Agatston units measured by electron beam CT scanning
* Written informed consent
* Negative serum pregnancy test if appropriate
* Expect to comply with protocol procedures and schedule

Exclusion Criteria:

* Unstable angina pectoris
* Severe congestive heart failure
* Severe obstructive pulmonary disease requiring supplemental oxygen
* Severe liver dysfunction
* Severe malnutrition
* Severe hyperparathyroidism
* Known HIV
* Active malignancy for which the subject is receiving chemotherapy or radiation
* Planned renal transplant within the next year
* Clinical evidence of calciphylaxis or recent history of hypercalcemia
* History of obstructed bowels
* Hypersensitivity to any of the components of the study medication
* History of swallowing disorders
* Weight > 300 pounds
* Any condition which makes patient participation not in the patient's best interest

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2005-01; Primary Completion 2006-12 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
electron-beam CT coronary artery calcification AGATSTON score | change at 12 mo from baseline

SECONDARY OUTCOMES:
serum phosphorus | Days 30-365
calcium x phosphorus product | Days 30-365

CONTACTS AND LOCATIONS:
Overall Officials: Wajeh Y Qunibi, M.D., Study Chair — The University of Texas Health Science Center at San Antonio
Locations (1):
- University of Texas Health Sciences Center, San Antonio, Texas, United States

REFERENCES:
- [Background] Chertow GM, Burke SK, Raggi P; Treat to Goal Working Group. Sevelamer attenuates the progression of coronary and aortic calcification in hemodialysis patients. Kidney Int. 2002 Jul;62(1):245-52. doi: 10.1046/j.1523-1755.2002.00434.x. PMID 12081584
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086
- [Derived] Qunibi W, Moustafa M, Muenz LR, He DY, Kessler PD, Diaz-Buxo JA, Budoff M; CARE-2 Investigators. A 1-year randomized trial of calcium acetate versus sevelamer on progression of coronary artery calcification in hemodialysis patients with comparable lipid control: the Calcium Acetate Renagel Evaluation-2 (CARE-2) study. Am J Kidney Dis. 2008 Jun;51(6):952-65. doi: 10.1053/j.ajkd.2008.02.298. Epub 2008 Apr 18. PMID 18423809